CLINICAL TRIAL: NCT02693509
Title: Get With The Guidelines-Heart Failure Registry
Status: Recruiting | Type: Observational
Sponsor: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: GWTG01
Record Dates: First submitted 2013-04-08; First posted 2016-02-26 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: GWTG Heart Failure program — Evidence based guideline recommended therapies and counseling prior to hospital discharge

SUMMARY:
Get With The Guidelines-Heart Failure is designed to improve the quality of care in patients hospitalized with heart failure. The program aims to help ensure that eligible patients are initiated on guideline recommended therapies and receive appropriate counseling prior to hospital discharge.

DETAILED DESCRIPTION:
Get With The Guidelines-Heart Failure was initiated in 2005 with over 500 U.S. hospitals participating is designed to improve the quality of care in patients hospitalized with heart failure. The program aims to help ensure that eligible patients are initiated on guideline recommended therapies and receive appropriate counseling prior to hospital discharge.

Peer-reviewed research(with over 35 manuscripts) has demonstrated that through participating in Get With The Guidelines-Heart Failure, hospitals will provide equitable care (regardless of race, ethnicity, age, or gender), the importance of scheduled physician follow-up after heart failure hospital discharge, the value in device-support as necessary for the acute heart failure patient, and many other significant findings.

Achievement measures tracked through Get With The Guidelines-Heart Failure:

* Angiotensin converting enzyme inhibitor (ACEI) and angiotensin receptor blocker (ARB) at discharge
* Evidence-based specific beta blockers
* Measure left ventricular function
* Post-discharge appointment for heart failure patients

Quality Measures tracked through Get With The Guidelines-Heart Failure:

* Mineralocorticoid receptor antagonist at discharge
* Aldosterone antagonist at discharge
* Anticoagulation for atrial fibrillation
* Hydralazine nitrate at discharge
* DVT prophylaxis
* CRT-D or CRT-P placed or prescribed at discharge
* ICD counseling, or ICD placed or prescribed at discharge
* Influenza vaccination during flu season
* Pneumococcal vaccination
* Follow-up visit within 7 days or less
* Lab monitoring follow-up
* SGLT-2 inhibitor at discharge
* Defect-free care for quadruple therapy medication for patients with heart failure with reduced ejection fraction
* Direct-acting oral anticoagulant at discharge for non-valvular atrial fibrillation or atrial flutter patients

Additional measures collected by Get With The Guidelines-Heart Failure can be viewed at: http://www.heart.org/idc/groups/heart-public/@wcm/@private/@hcm/@gwtg/documents/downloadable/ucm_310967.pdf

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with congestive heart failure.

Exclusion Criteria:

* Patients who do not have congestive heart failure,
* Patients under age of 18,
* Patients not admitted as inpatients.

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study populations is primary diagnosis or secondary diagnosis of heart failure
Sampling Method: Probability Sample
Enrollment: 128026 (Estimated)
Dates: Start 2005-01; Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
30 day readmission rate | 30 days post discharge from hospital
  Percent of index encounters where there is a readmission within 30 days
60 day readmission rate | 60 days post discharge from hospital
  Percent of index encounters where there is a readmission within 60 days
90 day readmission rate | 90 days post discharge from hospital
  Percent of index encounters where there is a readmission within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Javed Butler, MD, Study Director — American Heart Association
Locations (1):
- Amy Bennett, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] American Academy of Family Physicians; American Academy of Hospice and Palliative Medicine; American Nurses Association; American Society of Health-System Pharmacists; Heart Rhythm Society; Society of Hospital Medicine; Bonow RO, Ganiats TG, Beam CT, Blake K, Casey DE Jr, Goodlin SJ, Grady KL, Hundley RF, Jessup M, Lynn TE, Masoudi FA, Nilasena D, Pina IL, Rockswold PD, Sadwin LB, Sikkema JD, Sincak CA, Spertus J, Torcson PJ, Torres E, Williams MV, Wong JB; ACCF/AHA Task Force on Performance Measures; Peterson ED, Masoudi FA, DeLong E, Erwin JP 3rd, Fonarow GC, Goff DC Jr, Grady KL, Green LA, Heidenreich PA, Jenkins KJ, Loth A, Shahian DM. ACCF/AHA/AMA-PCPI 2011 performance measures for adults with heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Performance Measures and the American Medical Association-Physician Consortium for Performance Improvement. J Am Coll Cardiol. 2012 May 15;59(20):1812-32. doi: 10.1016/j.jacc.2012.03.013. Epub 2012 Apr 23. No abstract available. PMID 22534627
- [Derived] Rao VN, Mentz RJ, Coniglio AC, Kelsey MD, Fudim M, Fonarow GC, Matsouaka RA, DeVore AD, Caughey MC. Neighborhood Socioeconomic Disadvantage and Hospitalized Heart Failure Outcomes in the American Heart Association Get With The Guidelines-Heart Failure Registry. Circ Heart Fail. 2022 Nov;15(11):e009353. doi: 10.1161/CIRCHEARTFAILURE.121.009353. Epub 2022 Nov 15. PMID 36378758